CLINICAL TRIAL: NCT04634279
Title: Competitive Revision for Improving Access and Treatment for Co-occurring Opioid Use Disorders and Mental Illness
Brief Title: Competitive Revision for CLARO: Collaboration Leading to Addiction Treatment and Recovery From Other Stresses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of New Mexico (Other); Boston Medical Center (Other); Hidalgo Medical Services (Unknown); First Choice Community Healthcare (Unknown); Stanford University (Other); University of Pittsburgh (Other); Olive View-UCLA Education & Research Institute (Other); Saint John's Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3UF1MH121954-01S1 (NIH); 3UF1MH121954-01S1 (NIH)
Record Dates: First submitted 2020-11-02; First posted 2020-11-18 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Opioid-use Disorder; Addiction; Depression; Post Traumatic Stress Disorder; Suicidal Ideation
Keywords: Collaborative care; Problem Solving Therapy; Written Exposure Therapy; Medication for addiction treatment; Addiction; Opioid use disorder; Suicide prevention; Overdose prevention
MeSH Terms: conditions — Opioid-Related Disorders; Behavior, Addictive; Depression; Stress Disorders, Post-Traumatic; Suicidal Ideation; Suicide Prevention

STUDY DESIGN:
Intervention Model Description: Two-arm randomized control trial (RCT) where participants are randomly assigned to intervention or control.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Collaborative Care Plus (Experimental): Intervention is administered to patients in this arm. Care to be delivered via collaborative care. The supplement intervention adds family involvement in care and Caring Contacts, a suicide prevention method.
  Interventions: Behavioral: Collaborative care Plus
- Control (No Intervention): Patients in this arm will receive enhanced usual care.

INTERVENTIONS:
Behavioral: Collaborative care Plus — Collaborative care consists of a team of providers that includes a care coordinator, a primary care provider (PCP) and a behavioral health consultant (BHC), who provide evidence- and measurement-based care to a panel of patients using a clinical registry. In this model, the CC team also includes a behavioral health psychotherapist (BHP) who consults on a regular basis but does not deliver direct care. In the Collaborative Care Plus condition, the care coordinator involves family in care, teaches family about naloxone use, and provides Caring Contacts, a suicide prevention method, to patients.
  Arms: Collaborative Care Plus

SUMMARY:
The purpose of this study is to develop and then test an enhanced version of the parent study's collaborative care intervention for co-occurring disorders (CC-COD) to reduce the risk of suicide and overdose among individuals with opioid use disorder (OUD) in combination with PTSD/depression. The parent study is CLARO, Collaboration Leading to Addiction Treatment and Recovery from Other Stresses (NCT04559893).

DETAILED DESCRIPTION:
People with OUD co-occurring with depression or PTSD (COD) may not seek out treatment for their substance use or mental health issues, but they do visit their primary care provider. However, because providers generally lack specialized training in substance use and mental illness and are focused on the immediate reason for the visit, patients' substance use and mental disorders often go unrecognized and untreated. This missed opportunity can have lethal consequences. Individuals with COD are at higher risk of dying from suicide or overdose than individuals with mental illness or OUD alone. The parent study (NCT04559893) will provide a definitive answer as to whether collaborative care (CC) improves access, quality, and outcomes of care for individuals with COD. While a primary goal is to improve access to and retention in medication treatment for OUD (MOUD) (which is linked to decreased mortality and overdose risk), the interventions CC-COD supports do not proactively address suicide or overdose risk, an important limitation. In addition, CC-COD does not include families in the patient's care. The investigators address these limitations and tackle the public health crisis of increasing deaths from suicide and overdose with this study. Because family members can play an important role in a patient's decision to engage with treatment and in overdose and suicide prevention, the study team investigates family members' views and use this information to strengthen CC-COD. This revision will develop and then test the incremental effectiveness of three additional CC-COD components. Care coordinators will (1) educate family members about MOUD with the goal of increasing patient retention in treatment; (2) train family members and the patient to administer naloxone and on how to reduce overdose risk behaviors; and (3) implement Caring Contacts, a suicide prevention intervention that sends compassionate mailed or text messages to individuals to decrease social isolation and reduce suicide risk.

ELIGIBILITY:
Inclusion Criteria:

* 18 and older
* Receiving primary care at one of the participating clinical sites
* Has OUD and one or more specific co-occurring behavioral health disorders (depression and PTSD)

Exclusion Criteria:

* Under 18
* Does not speak English or Spanish
* Unable to consent
* Receiving both MOUD and psychotropic medication from a provider outside of the primary care health system at which the patient is enrolled.
* Not receiving primary care at one of the participating clinical sites

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2022-08-31 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2024-06-12 (Actual)

PRIMARY OUTCOMES:
MOUD continuity of care | Assessed over the first 180 days after study entry
  Max number of continuous (i.e., no breaks of more than 7 days) days the patient receives MOUD in the 180 days after study enrollment; obtained from electronic health record (EHR) or from the Prescription Drug Monitoring Program for the State of New Mexico

SECONDARY OUTCOMES:
Opioid overdose risk behaviors | Assessed over the previous 30 days at study entry and at 3 and 6 months after study entry
  Measured as a sum of ratings on 9 risk behaviors from Opioid Overdose Risk Assessment (score 0-36). A high score indicates high risk.
Suicide risk | Assessed over the previous 30 days at study entry and at 3 and 6 months after study entry
  Measured using Columbia Suicide Severity Rating Scales, classified into 6 levels (from no risk to suicide attempt)

OTHER OUTCOMES:
Demographics | Assessed at enrollment
  Sex, race, ethnicity, education level; assessed as moderators; obtained from patient interview
Alcohol use severity | Assessed over the previous 3 months at study entry
  10-item AUDIT for past 3 months; assessed as a covariate; obtained from patient interview
Pain levels | Assessed over the previous 7 days at enrollment and at 3 and 6 months
  Pain Intensity, Enjoyment of Life, General Activity (PEG) Pain Monitor for the past week; assessed as a covariate; obtained from patient interview
History of MOUD treatment | Asked about lifetime MOUD treatment; assessed at baseline
  Assessed as a covariate; obtained from patient interview
Current Major Depressive Disorder (MDD)/PTSD treatment | Assessed over the previous 30 days at study entry
  National Survey on Drug Use and Health (NSDUH) items; assessed as a covariate; obtained from patient interview
Prior experience with a care coordinator | Assessed over the previous 12 months at study entry
  Assessed as a covariate; obtained from patient interview
Interpersonal support | Asked about present state at time of measurement; assessed at enrollment
  Indicated by the patient identifying a support person with whom they interact and who does not have problematic opioid use;; obtained from patient interview
Homelessness | Assessed over the previous 3 months at study entry
  Homelessness Screening Clinical Reminder Tool and one item from the Government Performance and Results Act (GPRA) clarifying where individuals who are homeless are currently living; assessed as a mediator; obtained from patient interview. The study team constructed a single measure from the items described. They will not be analyzed separately as two different measures.
Legal involvement | Asked about lifetime legal involvement; assessed at baseline and at 3 and 6 months
  Items from the NSDUH and the Addiction Severity Index; assessed as a covariate; obtained from patient interview. The study team constructed a single measure from the items described. They will not be analyzed separately as two different measures.
Disability and impairment | Assessed over the previous 7 days at study entry
  3-item Sheehan Disability Scale; assessed as a covariate; obtained from patient interview
Rurality | Asked about present state at time of measurement; assessed at baseline
  Rural-Urban Commuting Area code associated with the participant's five-digit zip code; assessed as a moderator
Clinician (care coordinator) communication | Assessed over the previous 3 months at 3 months after study entry
  Agency for Healthcare Research and Quality (AHRQ) Consumer Assessment of Healthcare Providers and Systems survey items; assessed as a mediator; obtained from patient interview
Ability to access treatment quickly | Assessed over the previous 3 months at 3 months after study entry
  AHRQ Consumer Assessment of Healthcare Providers and Systems survey items; assessed as a mediator; obtained from patient interview
Satisfaction with treatment | Assessed over the previous 3 months at 3 months after study entry
  AHRQ Consumer Assessment of Healthcare Providers and Systems survey items; assessed as a mediator; obtained from patient interview
Patient-care coordinator working alliance | Assessed over the previous 3 months at 3 months after study entry
  Modified Working Alliance Inventory-General Practitioner (WAI-GP); assessed as a mediator; obtained from patient interview

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Watkins, MD, Principal Investigator — RAND; Miriam Komaromy, Principal Investigator — Boston Medical Center
Locations (12):
- United States (12):
  - Hubert Humphrey Comprehensive Health Center, Los Angeles, California
  - Providence Saint John's Health Center, Santa Monica, California
  - First Choice Community Healthcare - South Broadway Medical Center, Albuquerque, New Mexico
  - First Choice Community Healthcare - South Valley Medical/Dental Center, Albuquerque, New Mexico
  - First Choice - Alameda Medical Center, Albuquerque, New Mexico
  - First Choice Community Healthcare - North Valley Medical Center, Albuquerque, New Mexico
  - University of New Mexico Family Health Clinic, North Valley, Albuquerque, New Mexico
  - University of New Mexico Family Health Clinic, Southeast Heights, Albuquerque, New Mexico
  - First Choice Community Healthcare - Alamosa Medical Center, Albuquerque, New Mexico
  - First Choice Community Healthcare - Belen Medical Center, Belen, New Mexico
  - First Choice Community Healthcare - Edgewood Medical/Dental Center, Edgewood, New Mexico
  - First Choice Community Healthcare - Los Lunas Medical/Dental Center, Los Lunas, New Mexico

IPD SHARING:
Plan to Share IPD: Yes
Per National Institute of Mental Health (NIMH) funding requirements, study data must be uploaded to the NIMH National Data Archive (NDA) every six months once data collection begins. A universal subject identification, Global Unique Identifier, (GUID) will be generated for each participant. All raw data will be uploaded every six months to the NIMH NDA per their policies. Additionally, all analysis data sets used for manuscripts must be uploaded to the NIMH NDA, identified by GUID.
Time Frame: Every 6 months (January and July) following enrollment of the first patient. First submission expected July 2021. Submission will cease following sharing of final analysis data set for any specified outcomes publications.
Access Criteria: Per NIMH NDA policies
URL: https://nda.nih.gov/

REFERENCES:
- [Background] Fendrich M, Becker J, Hernandez-Meier J. Psychiatric symptoms and recent overdose among people who use heroin or other opioids: Results from a secondary analysis of an intervention study. Addict Behav Rep. 2019 Aug 6;10:100212. doi: 10.1016/j.abrep.2019.100212. eCollection 2019 Dec. PMID 31692644
- [Background] Ilgen MA, Bohnert AS, Ignacio RV, McCarthy JF, Valenstein MM, Kim HM, Blow FC. Psychiatric diagnoses and risk of suicide in veterans. Arch Gen Psychiatry. 2010 Nov;67(11):1152-8. doi: 10.1001/archgenpsychiatry.2010.129. PMID 21041616
- [Background] Jones CM, McCance-Katz EF. Co-occurring substance use and mental disorders among adults with opioid use disorder. Drug Alcohol Depend. 2019 Apr 1;197:78-82. doi: 10.1016/j.drugalcdep.2018.12.030. Epub 2019 Feb 14. PMID 30784952
- [Background] Moscicki EK, O'Carroll P, Rae DS, Locke BZ, Roy A, Regier DA. Suicide attempts in the Epidemiologic Catchment Area Study. Yale J Biol Med. 1988 May-Jun;61(3):259-68. PMID 3262956
- [Derived] Watkins KE, Osilla KC, McCullough CM, Griffin BA, Dopp AR, Becker K, Meredith LS, Carrejo V, Hindmarch GM, Mendon-Plasek S, Christensen J, Weir R, Kelly L, Pak L, Murray-Krezan C, Tarhuni L, Crowley C, Bilder A, Kalmin MM, Schoenbaum M, Komaromy M. Collaborative Care for Opioid Use Disorder and Mental Illness: The CLARO Randomized Clinical Trial. JAMA Intern Med. 2025 Dec 29:e257036. doi: 10.1001/jamainternmed.2025.7036. Online ahead of print. PMID 41460640
- [Derived] Osilla KC, Dopp AR, Watkins KE, Ceballos V, Hurley B, Meredith LS, Leamon I, Jacobsohn V, Komaromy M. Collaboration Leading to Addiction Treatment and Recovery from Other Stresses (CLARO): process of adapting collaborative care for co-occurring opioid use and mental disorders. Addict Sci Clin Pract. 2022 Apr 8;17(1):25. doi: 10.1186/s13722-022-00302-9. PMID 35395811